CLINICAL TRIAL: NCT06939400
Title: Study on Precision Photodynamic Therapy for Glioblastoma Multiforme Based on Metaverse and Yellow Fluorescence
Brief Title: Photodynamic Therapy for Glioblastoma Multiforme Based on Metaverse and Yellow Fluorescence
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Hushaoshan, Head of neurosurgery department, Zhejiang Provincial People's Hospital
Other Study IDs: KY2024208
Record Dates: First submitted 2025-02-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: Glioblastoma Multiforme; photodynamic therapy; metaverse; yellow fluorescence
MeSH Terms: conditions — Glioblastoma | interventions — Photochemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: GBM patients recevied traditional treatment options (including surgery combined with radiotherapy and chemotherapy)
  Interventions: Procedure: GBM patients recevied traditional treatment options
- Treatment: GBM patients recevied surgical combination photodynamic therapy
  Interventions: Procedure: Photodynamic therapy (PDT)

INTERVENTIONS:
Procedure: Photodynamic therapy (PDT) — GBM patients recevied surgical combination photodynamic therapy
  Other Names: Surgical combination photodynamic therapy
  Groups: Treatment
Procedure: GBM patients recevied traditional treatment options — GBM patients recevied traditional treatment options (including surgery combined with radiotherapy and chemotherapy)
  Groups: Control

SUMMARY:
GBM patients receiving PDT treatment (50 cases，surgery combined with photodynamic therapy) and traditional treatment (50 cases，traditional surgery) in our hospital and partner hospitals were collected. The prognosis was analyzed by comparing with the control group from multiple perspectives such as image evaluation, imaging effect, Karnofsky score, median survival time and survival rate.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed primary focal GBM; Recurrent GBM(single or satellite lesions); Multiple (multiple germinal centers)GBM.

Exclusion Criteria:

* Photosensitizer allergy.

  * Severe coagulation disorder.

    * Patients with severe cardiovascular and cerebrovascular diseases, especially patients in the acute stage.

      * Multiple organ failure, end-stage patients. ⑤ Pregnant women: Photofrin is considered a class C pregnancy risk (toxic, non-teratogenic) drug with non-dialysis properties.

Non-gbm diagnosis: Patients with other types of brain tumors or diseases. 7 Do not agree to informed consent: patients who are unwilling to sign informed consent or do not agree to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GBM patients recevied traditional treatment options (including surgery combined with radiotherapy and chemotherapy) or PDT treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment of Surgical combination Photodyanmic therapy | From June 2025 to June 2027

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No